CLINICAL TRIAL: NCT02822664
Title: Analysis of Cerebral Correlates of Pedophilia With Neuroimaging Techniques
Acronym: PCNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2008-535
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2016-06

CONDITIONS: Pedophilia
Keywords: Brain, pedophilia, neuroimaging
MeSH Terms: conditions — Pedophilia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pedophiles patients (Other): Adults diagnosed with pedophilia
  Interventions: Behavioral: Pedophiles patients; Device: PET/MRI
- Healthy subjects (Other): Healhy subjects (not diagnosed with pedophilia)
  Interventions: Behavioral: Healthy subjects; Device: PET/MRI

INTERVENTIONS:
Behavioral: Pedophiles patients — cerebral MRI and/or cerebral PET imaging
  Arms: Pedophiles patients
Behavioral: Healthy subjects — cerebral MRI and/or cerebral PET imaging
  Arms: Healthy subjects
Device: PET/MRI

SUMMARY:
The main objective is to identify cerebral correlated of pedophilia using neuroimaging techniques.

ELIGIBILITY:
Inclusion Criteria (for patients):

* Diagnosis of pedophilia
* Male
* Age between 18 and 65
* Informed consent signed

Inclusion Criteria (for healthy patients):

* Male
* Age between 18 and 65
* Informed consent signed

Exclusion Criteria (for patients):

* IQ <70
* Ongoing treatment with cyprostrerone acetate or GnRH agonist or antidepressant treatment (5HT reuptake inhibitor)
* Ongoing detention

Exclusion Criteria (for healthy patients):

* psychiatric disorders
* IQ<70
* Sexual disorders

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
BOLD contrast signal | 3 months
  Assesment of physiological measurements by Magnetic resonance imaging (MRI)
Local cerebral blood flow | 3 months
  Assesment of physiological measurements by Positron Emission Tomography (PET)

CONTACTS AND LOCATIONS:
Overall Officials: Michel PUGEAT, Prof, Principal Investigator — Hospices Civils de Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fonteille V, Redoute J, Lamothe P, Straub D, Lavenne F, Le Bars D, Raverot V, Moulier V, Marchand JJ, Vittoz A, Leriche C, Pugeat M, Stoleru S. Brain processing of pictures of children in men with pedophilic disorder: A positron emission tomography study. Neuroimage Clin. 2019;21:101647. doi: 10.1016/j.nicl.2018.101647. Epub 2018 Dec 24. PMID 30612938